CLINICAL TRIAL: NCT00204893
Title: Evaluation of the Ocular Safety of Calcium Formate in Normal, Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Nephro-Tech 1, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2003-297
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — formic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label (Experimental): Each participant will be treated with three 3900 mg doses of calcium formate on each study day (i.e., days 1-14).
  Interventions: Drug: calcium formate

INTERVENTIONS:
Drug: calcium formate — Calcium formate - Each uncoated white tablet will contain 650 mg of calcium formate, (equivalent to 200 mg elemental calcium). Nephro-Tech, LLC, will formulate and provide the calcium formate tablets for the study.

SUMMARY:
This is a Phase I, single center, open-label study of the dietary supplement calcium formate in normal, healthy female subjects. The purpose of the study is to determine whether daily use of calcium formate is safe and whether it accumulates in the eye.

DETAILED DESCRIPTION:
This is a Phase I, single center, open-label study of the dietary supplement calcium formate in normal, healthy female subjects. The purpose of the study is to determine whether daily use of calcium formate is safe and whether it accumulates in the eye.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females

Exclusion Criteria:

* no ocular diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Vision Testing (refraction) over baseline | Up to 15 days
  Participants will be refracted at baseline and the resultant lens correction will be used for testing visual acuity at all subsequent visits. If a participant's visual acuity drops 10 letters or more at any visit, the participant will be re-refracted and the visual acuity will be tested again with the new lens correction in place.
Change in Serum Formate Levels over baseline | Up to 15 days
  To test for accumulation of formate, morning blood samples for determination of formate will be obtained at screening, prior to administration of the first dose of calcium formate on Study Days 1, 2, 3, and 8 and on day 15. Blood samples for determination of formate will also be obtained approximately 40-60 minutes after ingestion of the second dose on Study Days 1, 2 and 3.

SECONDARY OUTCOMES:
Change in Visual Acuity over baseline | Up to 15 days
  Based on retroilluminated Chart R from Ferris-Bailey Early Treatment Diabetic Retinopathy Study (ETDRS) distance visual acuity chart set.
Change in 100 Hue Vision Testing results over baseline | Up to 15 days
  The FM-100 Hue test will be utilized to assess color vision at baseline and at the conclusion of the study. This test requires the arrangement of 100 discs of varying hues in an orderly sequence. The test requires 15 minutes to complete and is noninvasive. The test is scored by a computer.
Change in ERG/VEP over baseline | Up to 15 days
  Change in electroretinography (ERG) and visual-evoked potential will be monitored over baseline.
Change in Visual Fields over baseline | Up to 15 days
  Automated standardized Humphrey 24-2 visual fields will be performed using the SITA (Swedish Interactive Threshold Algorithm) protocol. This test is standard of care for the assessment and follow-up of optic nerve disorders such as glaucoma or optic neuropathy. It will be performed in the customary manner for evaluation of mean defect.
Fundus Photography | Up to 15 days
  Stereoscopic color fundus photographs of both eyes will be taken with a 30 degree fundus camera at baseline, at day 2 and day 8 of study tablet administration 40-60 minutes after the second dose, and at study completion (day 15), early termination, or if a vision drop or AE occurs. These will be compared individually for changes including macular edema, retinal or optic nerve abnormalities or other abnormalities occurring from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Altaweel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Altaweel MM, Hanzlik RP, Ver Hoeve JN, Eells J, Zhang B. Ocular and systemic safety evaluation of calcium formate as a dietary supplement. J Ocul Pharmacol Ther. 2009 Jun;25(3):223-30. doi: 10.1089/jop.2008.0128. PMID 19456257